CLINICAL TRIAL: NCT04973046
Title: Tissue Oxygen Saturation During Gastric Tube Reconstruction With Cervical Anastomosis for Esophagectomy
Brief Title: Tissue Oxygen Saturation for Esophagectomy
Status: Completed | Type: Observational
Sponsor: Shizuoka Cancer Center (Other)
Responsible Party: Principal Investigator, Kenjiro Ishii, Principal Investigator, Shizuoka Cancer Center
Other Study IDs: ShizuokaCC rSO2
Record Dates: First submitted 2021-07-03; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Esophageal Neoplasms; Esophagostomy Complication; Anastomotic Leak; Oxygen Deficiency
Keywords: Esophagectomy, Tissue oxygen saturation, Gastric tube, Anastomotic leakage
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak; Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tissue oxygen saturation monitoring was a useful indicator of blood flow insufficiency in the gastric tube leading to anastomotic leakage during radical esophagectomy.

DETAILED DESCRIPTION:
One cause of anastomotic leakage after radical esophagectomy is blood flow insufficiency at the cervical anastomosis site. .

Eighteen patients, who underwent radical esophagectomy with gastric tube reconstruction, were studied. The regional tissue oxygen saturation (rSO2) was measured at the tip (point pre 0) and 2, 4, and 6 cm on the anal side of the tip (point pre 1, pre 2, and pre 3, respectively) before the gastric tube was raised to the cervical site through the retrosternal route. After that, rSO2 was measured at the tip, 2 and 4 cm on the anal side of the tip (points post 0, post 1, and post 2), the actual anastomotic site (point AN), and the chest skin as an indicator of whole-body oxygenation . The relationship between rSO2 scores and the rate of anastomotic leakage was determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent esophagectomy with gastric tube reconstruction from November 2020 to March 2021.

Exclusion Criteria:

* Patients who underwent esophagectomy with jejunum or colon reconstruction. patients who underwent two-stage operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective study performed at the Shizuoka Cancer Center between November 2020 and March 2021. All 18 patients who underwent esophagectomy with gastric tube reconstruction were enrolled in the study
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The tissue oxygen saturation score of gastric tube during esophagectomy | During surgery
  We measured the tissue oxygen saturation (0% - 99%) of several parts of gastric tube during esophagectomy with a use of tissue saturation monitor ''toccare''.

SECONDARY OUTCOMES:
The rate of anastomotic leakage | 1month after surgery
  We investigated the rate of anastomotic leakage in the cervical site (0% - 100%).

CONTACTS AND LOCATIONS:
Locations (1):
- Shizuoka cancer center, Nagaizumicho, Suntogun, Japan